CLINICAL TRIAL: NCT00896454
Title: A Single-arm, Multicenter, Proof-of-concept Study of Denosumab in the Treatment of Hypercalcemia of Malignancy in Subjects With Elevated Serum Calcium Despite Recent Treatment With IV Bisphosphonates
Brief Title: Study of Denosumab in the Treatment of Hypercalcemia of Malignancy in Subjects With Elevated Serum Calcium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20070315
Record Dates: First submitted 2009-05-07; First posted 2009-05-11 (Estimated); Results first posted 2015-01-01 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Breast Cancer; Hypercalcemia of Malignancy; Colon Cancer; Endocrine Cancer; Head and Neck Cancer; Kidney Cancer; Lung Cancer; Lymphoma; Metastatic Cancer; Multiple Myeloma; Parathyroid Neoplasms; Renal Cancer; Thyroid Cancer; Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma; Non-Small Cell Lung Cancer
Keywords: hypercalcemia; calcium; bisphosphonates; denosumab; amgen; malignancy; 20070315; HMC; oncology; hematology
MeSH Terms: conditions — Breast Neoplasms; Humoral Hypercalcemia Of Malignancy; Colonic Neoplasms; Endocrine Gland Neoplasms; Head and Neck Neoplasms; Kidney Neoplasms; Lung Neoplasms; Lymphoma; Neoplasm Metastasis; Multiple Myeloma; Parathyroid Neoplasms; Thyroid Neoplasms; Hodgkin Disease; Lymphoma, Non-Hodgkin; Carcinoma, Non-Small-Cell Lung; Hypercalcemia; Neoplasms | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- denosumab (Experimental): Eligible subjects will receive denosumab at a dose of 120 mg subcutaneously (SC) every 4 weeks (Q4W) with a loading dose of 120 mg SC on study days 8 and 15.
  Interventions: Drug: denosumab

INTERVENTIONS:
Drug: denosumab — 120 mg subcutaneously (SC) every 4 weeks with a loading dose of 120 mg SC on study days 8 and 15.

SUMMARY:
The purpose of this study is to determine the potential of denosumab to treat Hypercalcemia of Malignancy in patients with elevated serum calcium who do not respond to recent treatment with intravenous bisphosphonates by lowering corrected serum calcium </= 11.5 mg/dL (2.9 millimoles /L) by day 10.

ELIGIBILITY:
Inclusion Criteria:

* Hypercalcemia of Malignancy (HCM) as defined as documented histologically or cytologically confirmed cancer and a corrected serum calcium (CSC) > 12.5 mg/dL (3.1 millimoles /L) at screening by local laboratory
* Last IV bisphosphonate treatment must be >/= to 7 days and </= to 30 days before the screening corrected serum calcium
* Adults (>/=18 years)
* Adequate organ function as defined by the following criteria:
* serum aspartate aminotransferase (AST) </= 5 x upper limit of normal (ULN)
* serum alanine aminotransferase (ALT) </= 5 x upper limit of normal
* serum total bilirubin </= 2 x upper limit of normal

Exclusion Criteria:

* Evidence of benign hyperparathyroidism, hyperthyroidism, adrenal insufficiency, vitamin D intoxication, milk alkali syndrome, sarcoidosis, or other granulomatous disease
* Receiving dialysis for renal failure
* Treatment with thiazides, calcitonin, mithramycin, or gallium nitrate within their window of expected therapeutic effect (as determined by the physician) prior to the date of the screening CSC
* Treatment with cinacalcet within 4 weeks prior to the date of the screening CSC
* Thirty days or less since receiving an investigational product (other than denosumab) or device (ie, does not have marketing authorization; thalidomide use is allowed) in another clinical study
* Known sensitivity to any of the products to be administered during the study (eg, mammalian derived products)
* Female subject is pregnant or breast feeding, or planning to become pregnant within 7 months after the end of treatment
* Female subject of childbearing potential is not willing to use 2 highly effective methods of contraception during treatment and for 7 months after the end of treatment
* Subject will not be available for follow-up assessment.
* Any organic or psychiatric disorder that, in the opinion of the investigator, might prevent the subject from completing the study or interfere with the interpretation of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-11-16 (Actual); Primary Completion 2012-09-13 (Actual); Study Completion 2013-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (24):
- United States (12):
  - Research Site, Encinitas, California
  - Research Site, New Haven, Connecticut
  - Research Site, Salisbury, Maryland
  - Research Site, Dearborn, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Omaha, Nebraska
  - Research Site, New York, New York
  - Research Site, Syracuse, New York
  - Research Site, The Bronx, New York
  - Research Site, Durham, North Carolina
  - Research Site, Goldsboro, North Carolina
  - Research Site, Houston, Texas
- Canada (2):
  - Research Site, QuÃ©bec, Quebec
  - Research Site, Québec, Quebec
- France (4):
  - Research Site, Limoges
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Villejuif
- Italy (5):
  - Research Site, Bologna
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Roma
- Research Site, Warsaw, Poland

REFERENCES:
- [Derived] Hu MI, Glezerman I, Leboulleux S, Insogna K, Gucalp R, Misiorowski W, Yu B, Ying W, Jain RK. Denosumab for patients with persistent or relapsed hypercalcemia of malignancy despite recent bisphosphonate treatment. J Natl Cancer Inst. 2013 Sep 18;105(18):1417-20. doi: 10.1093/jnci/djt225. Epub 2013 Aug 29. PMID 23990665
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient was enrolled on 16 November 2009 and the last patient enrolled on 02 July 2012. Data are reported as of the primary analysis cut-off date of 13 September 2012.
Groups:
- Denosumab: Participants received denosumab at a dose of 120 mg subcutaneously (SC) every 4 weeks (Q4W) with a loading dose of 120 mg SC on study Days 8 and 15.
Period: Overall Study
Arm/Group | Denosumab
Started | 33
Completed | 0
Not Completed | 33
Not completed — Death | 10
Not completed — Adverse Event | 8
Not completed — Disease Progression | 5
Not completed — Other | 4
Not completed — Requirement for alternative therapy | 3
Not completed — Ongoing in study | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Denosumab
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 21
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 23
  Black or African American | 7
  Hispanic or Latino | 1
  Asian | 1
  Other | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Scale used to assess how a patient's disease is progressing, how the disease affects the daily living abilities of the patient: 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory, able to carry out work of a light nature; 2 = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self care, confined to a bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  participants
    0 | 1
    1 | 7
    2 | 14
    3 | 8
    4 | 3
Primary Tumor Type [Number; unit: participants]
  Bladder | 1
  Breast | 6
  Head and neck | 2
  Liver | 1
  Neuroendocrine/carcinoid | 4
  Non-hodgkin's | 2
  Non-small cell lung cancer | 3
  Ovarian | 1
  Renal | 3
  Small cell lung cancer | 1
  Soft tissue sarcoma | 1
  Unknown (primary tumor) | 1
  Multiple myeloma | 3
  Chronic lymphocytic leukemia | 2
  IGG kappa multiple myeloma | 1
  Myeloma | 1
Time from initial cancer diagnosis to enrollment [Mean (Standard Deviation); unit: months] | 56.9 (68.8)
Presence of metastatic disease at enrollment [Number; unit: participants]
  Yes | 30
  No | 3
Presence of bone metastatic disease at enrollment [Number; unit: participants]
  Yes | 13
  No | 20
Baseline Hypercalcemia of Malignancy (HCM) Symptoms [Number; unit: participants] — Participants may have had more than one symptom
  participants
    Fatigue | 9
    Anorexia | 5
    Nausea | 4
    Depressed level of consciousness | 2
    Vomiting | 2
    Dry mouth | 1
    Constipation | 4
    Lethargy | 4
    Confusion | 3
    Polyuria | 2
    Abdominal pain | 1
    Decreased mental acuity | 1
    Dyspnea | 1
    General weakness | 1
    Insomnolence | 1
    Light headedness (dizziness) | 1
    Listlessness/muscle weakness | 1
    Polyuro-polydipsic syndrome | 1
    Psychomotor retardation | 1
    Retching | 1
    Urinary frequency | 1
    Weight loss | 1
Calcium (corrected) [Mean (Standard Deviation); unit: mg/dL] | 13.89 (1.27)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Response Within 10 Days of First Dose of Denosumab
Description: Response is defined as corrected serum calcium (CSC) ≤ 11.5 mg/dL, within 10 days after the first dose of denosumab. For all CSC values, if albumin was < 4 g/dL, the following formula was used to calculate CSC: CSC = Total serum calcium [mg/dL] + (0.8 x (4 - serum albumin [g/dL]))
Time Frame: 10 days
Population: Response Analysis Subset including all participants who received at least 1 dose of denosumab and had a screening CSC (from local lab) > 12.5 mg/dL (3.1 mmol/L).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Denosumab
Number analyzed (Participants) | 33
percentage of participants | 63.6 [45.1 to 79.6]

2. Secondary Outcome: Percentage of Participants With a Response by Visit
Description: as for outcome 1
Time Frame: Days 2, 4, 8, 10, 15, 19, 23, 29, 36, 43, 50 and 57
Population: Response Analysis Subset
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Denosumab
Number analyzed (Participants) | 33
percentage of participants
  By Day 2 | 9.1 [1.9 to 24.3]
  By Day 4 | 24.2 [11.1 to 42.3]
  By Day 8 | 48.5 [30.8 to 66.5]
  By Day 10 | 63.6 [45.1 to 79.6]
  By Day 15 | 63.6 [45.1 to 79.6]
  By Day 19 | 69.7 [51.3 to 84.4]
  By Day 23 | 69.7 [51.3 to 84.4]
  By Day 29 | 69.7 [51.3 to 84.4]
  By Day 36 | 69.7 [51.3 to 84.4]
  By Day 43 | 69.7 [51.3 to 84.4]
  By Day 50 | 69.7 [51.3 to 84.4]
  By Day 57 | 69.7 [51.3 to 84.4]

3. Secondary Outcome: Percentage of Participants With a Complete Response by Visit
Description: Response is defined as corrected serum calcium (CSC) ≤ 10.8 mg/dL (2.7 mmol/L). For all CSC values, if albumin was < 4 g/dL, the following formula was used to calculate CSC: CSC = Total serum calcium [mg/dL] + (0.8 x (4 - serum albumin [g/dL])).
Time Frame: Days 2, 4, 8, 10, 15, 19, 23, 29, 36, 43, 50 and 57
Population: Response Analysis Subset
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Denosumab
Number analyzed (Participants) | 33
percentage of participants
  By Day 2 | 3.0 [0.1 to 15.8]
  By Day 4 | 15.2 [5.1 to 31.9]
  By Day 8 | 27.3 [13.3 to 45.5]
  By Day 10 | 36.4 [20.4 to 54.9]
  By Day 15 | 45.5 [28.1 to 63.6]
  By Day 19 | 45.5 [28.1 to 63.6]
  By Day 23 | 51.5 [33.5 to 69.2]
  By Day 29 | 51.5 [33.5 to 69.2]
  By Day 36 | 60.6 [42.1 to 77.1]
  By Day 43 | 63.6 [45.1 to 79.6]
  By Day 50 | 63.6 [45.1 to 79.6]
  By Day 57 | 63.6 [45.1 to 79.6]

4. Secondary Outcome: Time to Response
Description: Time to Response was defined as the time period from study Day 1 to the first time post-baseline corrected serum calcium (CSC) ≤ 11.5 mg/dL. Participants were censored on the last CSC assessment day if no response was observed. If there was no post-baseline CSC assessment, time to response was censored on study Day 1.
  Time to response was analyzed using Kaplan-Meier methods.
Time Frame: From Day 1 until the end of study date or primary data cutoff date (13 September 2012), whichever occured first; median time on study was 1.8 months.
Population: Response Analysis Subset
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Denosumab
Number analyzed (Participants) | 33
days | 9.0 [5.00 to 19.00]

5. Secondary Outcome: Time to Complete Response
Description: Time to complete response was defined as the time period from study Day 1 to the first time post-baseline corrected serum calcium (CSC) was ≤ 10.8 mg/dL (2.7 mmol/L). Participants were censored on the last CSC assessment day if no complete response was observed. If there was no post-baseline CSC assessment, time to complete response was censored on study Day 1. Time to complete response was analyzed using Kaplan-Meier methods.
Time Frame: as for outcome 4
Population: Response Analysis Subset
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Denosumab
Number analyzed (Participants) | 33
days | 23.0 [11.00 to 43.00]

6. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the number of days from the first day of corrected serum calcium ≤ 11.5 mg/dL (2.9 millimoles/L) to the last day of corrected serum calcium ≤ 11.5 mg/dL. Participants were censored on the last CSC assessment day if their CSC level never reached > 11.5 mg/dL after the first response. If a participant had no CSC assessment after the first response, duration of response was set to zero and censored. Duration of response was summarized for participants who achieved a response using the Kaplan-Meier method.
Time Frame: as for outcome 4
Population: Participants with a response in the Response Analysis Subset
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Denosumab
Number analyzed (Participants) | 23
days | 104.0 [9.00 to NA] — Not estimable due to the low number of events

7. Secondary Outcome: Duration of Complete Response
Description: Duration of complete response is defined as the number of days from the first day of of corrected serum calcium ≤ 10.8 mg/dL (2.7 millimoles/L) to the last day of corrected serum calcium ≤ 10.8 mg/dL. Participants were censored on the last CSC assessment day if their CSC level never reached > 10.8 mg/dL after the complete response. If a participant had no CSC assessment after the complete response, duration of complete response was set to zero and censored. Duration of complete response was summarized for participants who achieved a complete response using the Kaplan-Meier method.
Time Frame: as for outcome 4
Population: Participants with a complete response in the Response Analysis Subset
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Denosumab
Number analyzed (Participants) | 21
days | 34.0 [1.00 to 134.00]

8. Secondary Outcome: Time to Relapse/Nonresponse of Hypercalcemia of Malignancy
Description: Time to relapse/nonresponse was defined as the number of days from study Day 1 until the last day of CSC ≤ 11.5 mg/dL for all particiipants with relapse after the first response. Participants were censored on the last CSC assessment day if their CSC level never reached > 11.5 mg/dL after first response. For participants who never achieved response, time to relapse/nonresponse was set to zero. Otherwise, if there was no post-baseline CSC assessment, time to relapse/nonresponse was censored on study Day 1. Time to relapse/nonresponse was estimated using the Kaplan-Meier method.
Time Frame: as for outcome 4
Population: Response Analysis Subset
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Denosumab
Number analyzed (Participants) | 33
days | 19.0 [5.00 to 114.00]

9. Secondary Outcome: Change From Baseline in Corrected Serum Calcium
Time Frame: Baseline and Days 2, 4, 8, 10, 15, 19, 23, 29, 36, 43, 50 and 57
Population: Efficacy Analysis Subset included all participants who received at least 1 dose of denosumab. n = Number of participants who had non-missing data at Baseline and the time point of interest.
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Denosumab
Number analyzed (Participants) | 33
mmol/L
  Change from Baseline to Day 2 (n = 32) | -0.13 [-0.31 to 0.09]
  Change from Baseline to Day 4 (n = 32) | -0.25 [-0.44 to -0.14]
  Change form Baseline to Day 8 (n = 27) | -0.43 [-0.73 to -0.20]
  Change from Baseline to Day 10 (n = 28) | -0.54 [-0.77 to -0.25]
  Change from Baseline to Day 15 (n = 24) | -0.51 [-0.89 to -0.15]
  Change from Baseline to Day 19 (n = 22) | -0.64 [-0.80 to -0.30]
  Change from Baseline to Day 23 (n = 21) | -0.60 [-0.85 to -0.40]
  Change from Baseline to Day 29 (n = 22) | -0.53 [-0.75 to -0.30]
  Change from Baseline to Day 36 (n = 20) | -0.61 [-0.84 to -0.15]
  Change from Baseline to Day 43 (n = 19) | -0.75 [-0.98 to -0.10]
  Change from Baseline to Day 50 (n = 15) | -0.83 [-1.03 to -0.20]
  Change from Baseline to Day 57 (n = 17) | -0.73 [-1.03 to -0.25]

ADVERSE EVENTS:
Time Frame: Median time on study was 1.8 months.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Denosumab 120 mg Q4W: Participants received denosumab at a dose of 120 mg subcutaneously (SC) every 4 weeks (Q4W) with a loading dose of 120 mg SC on study Days 8 and 15.
Arm/Group | Denosumab 120 mg Q4W
Serious Adverse Events (participants affected / at risk) | 29/33
Other Adverse Events (participants affected / at risk) | 26/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab 120 mg Q4W (N=33)
Anaemia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 2
Hypercalcaemia of malignancy (Endocrine disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Oesophageal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Septic shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urine output decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lethargy (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Renal tubular necrosis (Renal and urinary disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab 120 mg Q4W (N=33)
Anaemia (Blood and lymphatic system disorders) | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 7
Dry mouth (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 7
Asthenia (General disorders) | 2
Fatigue (General disorders) | 6
Oedema peripheral (General disorders) | 8
Pyrexia (General disorders) | 4
Pneumonia (Infections and infestations) | 3
Fall (Injury, poisoning and procedural complications) | 2
Haemoglobin decreased (Investigations) | 3
Weight decreased (Investigations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 7
Fluid overload (Metabolism and nutrition disorders) | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Depressed level of consciousness (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 8
Confusional state (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 3
Rash pruritic (Skin and subcutaneous tissue disorders) | 2
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.